CLINICAL TRIAL: NCT00688571
Title: Melody TPV Post-Market Surveillance Study
Brief Title: Melody Transcatheter Pulmonary Valve (TPV) Post-Market Surveillance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRC-CS-PMSS
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Heart Valve Diseases
Keywords: Pulmonary Valve; Congenital Heart Disease
MeSH Terms: conditions — Heart Valve Diseases; Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Melody TPV Implant (Experimental): Melody Transcatheter Pulmonary Valve implanted into a dysfunctional RV-PV conduit.
  Interventions: Device: Melody Transcatheter Pulmonary Valve

INTERVENTIONS:
Device: Melody Transcatheter Pulmonary Valve — Transcatheter valve implantation into a RV-PA conduit in patients with complex congenital heart defects where the conduit has become dysfunctional and where the patient needs intervention

SUMMARY:
This non-randomized, prospective, interventional observational multi-center study is designed to assess the long-term clinical performance of the Medtronic Melody™ Transcatheter Pulmonary Valve (TPV) in the post market environment over a period of five years after transcatheter implantation in patients with dysfunctional RVOT conduits. In addition, the quality of life of implanted subjects will be assessed over five years.

ELIGIBILITY:
Prospective subjects have complex congenital heart defects that have been palliated with RVOT conduits that have become dysfunctional and have a clinical indication for invasive intervention. Prospective subjects must meet all of following inclusion and exclusion criteria:

Inclusion Criteria:

* Age greater than or equal to 5 years of age
* Weight greater than or equal to 30 kilograms
* Existence of a full (circumferential) RVOT conduit that was equal to or greater than 16 mm in diameter when originally implanted
* Any of the following by transthoracic echocardiography

For patients in NYHA Classification II, III, or IV:

* Moderate (3+) or severe (4+) pulmonary regurgitation, or
* Mean RVOT gradient greater than or equal to 35 mmHg.

For patients in NYHA Classification I:

* Severe (4+) pulmonary regurgitation with RV dilatation or dysfunction, or
* Mean RVOT gradient greater than or equal to 40 mmHg.

Exclusion Criteria:

* Active endocarditis
* A major or progressive non-cardiac disease (e.g. liver failure, renal failure, cancer) that results in a life expectancy of less than one year
* Patient or - for patients who cannot legally give consent themselves- the guardian unwilling or unable to provide written informed consent or comply with follow-up requirements
* Obstruction of the central veins (including the superior and inferior vena cava, bilateral iliac veins) such that the delivery system cannot be advanced to the heart via transvenous approach from either femoral vein or internal jugular vein
* Known intravenous drug abuse

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2007-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Clinical Performance over five years. Freedom from the following events: * explant * reintervention * stent fracture * valve dysfunction * device or procedure related death | August 2014

SECONDARY OUTCOMES:
Procedural success | August 2014
Incidence of device and procedure related adverse events | August 2014
Hemodynamic Performance | August 2014

CONTACTS AND LOCATIONS:
Overall Officials: John Hess, Prof., Principal Investigator — Deutsches Herzzentrum München; Felix Berger, Prof., Principal Investigator — German Heart Institute; Lars Soendergaard, Dr., Principal Investigator — Rigshospitalet, Denmark; Maria Giulia Gagliardi, Dr., Principal Investigator — Ospedale Bambino Gesu Rome; Jose Suarez de Lezo, Dr., Principal Investigator — Hospital Reina Sofia Cordoba; Lee Benson, Dr., Principal Investigator — The Hospital for Sick Children; Maarten Witsenburg, Dr., Principal Investigator — Erasmus Medical Center
Locations (7):
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Rigshospitalet Copenhagen, Copenhagen, Denmark
- Germany (2):
  - Deutsches Herzzentrum Berlin, Berlin
  - Deutsches Herzzentrum München, München
- Hospital Bambino Gesu Roma, Rome, Italy
- Erasmus Medical Center, Rotterdam, Netherlands
- Hospital Reina Sofia, Córdoba, Spain

REFERENCES:
- [Derived] Armstrong AK, Berger F, Jones TK, Moore JW, Benson LN, Cheatham JP, Turner DR, Rhodes JF, Vincent JA, Zellers T, Lung TH, Eicken A, McElhinney DB. Association between patient age at implant and outcomes after transcatheter pulmonary valve replacement in the multicenter Melody valve trials. Catheter Cardiovasc Interv. 2019 Oct 1;94(4):607-617. doi: 10.1002/ccd.28454. Epub 2019 Aug 16. PMID 31419019
- [Derived] McElhinney DB, Benson LN, Eicken A, Kreutzer J, Padera RF, Zahn EM. Infective endocarditis after transcatheter pulmonary valve replacement using the Melody valve: combined results of 3 prospective North American and European studies. Circ Cardiovasc Interv. 2013 Jun;6(3):292-300. doi: 10.1161/CIRCINTERVENTIONS.112.000087. Epub 2013 Jun 4. PMID 23735475